CLINICAL TRIAL: NCT07113912
Title: Thoracic Mobilization Versus Counterforce Forearm Brace in Treatment of Lateral Elbow Tendinopathy (Randomized Control Trail)
Brief Title: Thoracic Mobilization Versus Counterforce Forearm Brace in Treatment of Lateral Elbow Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deraya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: physio 7 2025
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Lateral Elbow Tendinopathy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Received counterforce forearm brace and conventional therapy.
  Interventions: Device: counterforce forearm brace
- Control group (Active Comparator): Received thoracic mobilization and conventional therapy.
  Interventions: Procedure: thoracic immobilization

INTERVENTIONS:
Device: counterforce forearm brace — a flexible band that fits around the proximal forearm, applying pressure to underlying tissues during activity to potentially reduce acceleration forces and alleviate pain associated with conditions like lateral epicondylitis.
  Arms: Experimental group
Procedure: thoracic immobilization — the methods and devices used to restrict movement of the thoracic spine, which is the upper and middle part of the back.
  Arms: Control group

SUMMARY:
The study aim to compare the effect of thoracic mobilization versus counterforce forearm brace in treatment of LET.

Detailed Description:

Conditions: Lateral elbow tendinopathy Keywords: LET, Tennis elbow, Thoracic mobilization & counterforce forearm brace.

ELIGIBILITY:
Inclusion Criteria:

* Patients clinically diagnosed as lateral elbow tendinopathy.
* Positive clinical sign on the following: Cozen's test Mill's test and Maudsley's test
* Pain involving in age group of 18-55 years
* Patients complaining from unilateral elbow pain, more than 3 months

Exclusion Criteria:

* Previous Surgery or Intervention (e.g., tendon release, debridement, or joint replacement) in the affected shoulder/elbow are excluded
* Presence of systemic conditions affecting tendon healing like rheumatoid arthritis, diabetes, or other systemic diseases that impair tendon healing or exacerbate pain can confound results
* Severe Comorbidities Such as Severe cardiovascular, neurological, or musculoskeletal disorders

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 4 weeks
  consists of a 10 cm (or 100 mm) horizontal or vertical line, where 0 indicates no pain, and 10 (or 100 mm) represent the worst imaginable pain

CONTACTS AND LOCATIONS:
Locations (1):
- Deraya universuty, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided